CLINICAL TRIAL: NCT01733667
Title: A Prospective, Randomized, Multi-Center Evaluation of MediENT® Middle Turbinate Implant Versus MeroPack®, a Bioresorbable Nasal Dressing / Sinus Stent After Endoscopic Sinus Surgery
Acronym: MISTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ENTrigue Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSA2011-01
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Synechia
Keywords: synechia; Fess; sinus surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MediENT (Experimental): Right or left sinus cavity where MediENT will be place after randomization.
  Interventions: Device: MediENT
- MeroPack (Active Comparator): Right or left sinus cavity where MeroPack will be placed after randomization of MediENT is assigned.
  Interventions: Device: MeroPack

INTERVENTIONS:
Device: MediENT — MediENT will be assigned to either the right or left side and positioned between the turbinate and nasal wall of the side assigned. MeroPack will be place in between the turbinate and nasal wall of the side not assigned to MediENT
  Other Names: MeroPack
  Arms: MediENT
Device: MeroPack — MediENT will be assigned to either the right or left side and positioned between the turbinate and nasal wall of the side assigned. MeroPack will be place in between the turbinate and nasal wall of the side not assigned to MediENT
  Arms: MeroPack

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of MediENT to MeroPack after FESS.

DETAILED DESCRIPTION:
MediENT is designed to minimize lateralization of the middle turbinate, which can cause scarring and obstruction of key sinus openings after endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 18 and 65 years
2. Subject scheduled to undergo bilateral endoscopic sinus surgery
3. Subject signs IRB-approved informed consent form
4. Subject agrees to comply with all study-related procedures

Exclusion Criteria:

1. History of removal of one or both middle turbinates
2. Significant sinonasal polyps
3. Presence of marked septal asymmetry
4. Presence of significant concha bullosa, which requires surgical excision
5. Presence of non-viable tissue at the implantation site
6. Has an autoimmune disease, e.g., lupus, Graves' disease, myasthenia gravis, Wegener's granulomatosis
7. Known or suspected allergy to device components
8. Participating in another clinical trial which could affect the healing of the middle turbinate
9. Uncontrolled diabetes
10. Known or suspected use of illicit drugs
11. Known or suspected alcoholism
12. Other medical illness that could prevent follow-up or increase the risk of surgery
13. Pregnant or unwilling to take pregnancy prevention measures
14. Subject is currently using CPAP (Continuous Positive Airway Pressure) for sleep apnea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Miller synechia score at 8 weeks | 8 weeks post endoscopic sinus surgery
  Miller synechia score at 8 weeks (Number and degree of synechia present between middle turbinate and lateral nasal wall at 8 weeks judged by an independent evaluator)

SECONDARY OUTCOMES:
Miller Score at 4 & 8 weeks | 4 & 8 weeks post endoscopic sinus surgery
  * Miller synechia score at 4 weeks (Number and degree of synechia present between middle turbinate and lateral nasal wall at 4 weeks judged by an independent evaluator)
  * Total mean Miller score at 8 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Central California ENT Medical Group, Fresno, California
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Advanced ENT and Allergy, Louisville, Kentucky
  - ENT Associates of Texas, McKinney, Texas
  - Ear, Nose & Throat Clinics of San Antonio, San Antonio, Texas